CLINICAL TRIAL: NCT01565317
Title: Evaluation of the Effect of Intensive Diabetes Control Through Non-Surgical Intensive Lifestyle Modifications and Weight Reduction on Diabetic Peripheral Neuropathy
Brief Title: Evaluating the Effect of Diabetes Control Through Intensive Lifestyle Modifications on Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: NeuroMetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Osama Hamdy, Principal Investigator, Joslin Diabetes Center
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHS #2011-16
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Polyneuropathy; Weight Loss
MeSH Terms: conditions — Diabetic Neuropathies; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Treatment (Why WAIT) (Experimental): Weight Achievement and Intensive Treatment (Why WAIT) is a 12 -week multidisciplinary program for weight control and intensive diabetes management designed by the Joslin Diabetes Center for application in a multidisciplinary diabetes practice environment. Participants will be enrolled in a 12-week multidisciplinary intensive weight management including diet, exercise, behavioral and educational support. Participants will be enrolled in cohorts of 10-15 participants to encourage group interaction and support. Subjects will choose to come to the Joslin clinic every Tuesday or Wednesday evening for 2 hours. Participants will exercise for an hour and will attend a didactic session in the areas of nutrition, exercise and behavioral modifications.
  Interventions: Other: Weight Achievement and Intensive Treatment (Why WAIT)
- Control Group (No Intervention): Matched control group will be recruited from obese patients with diabetes followed at Joslin Clinic. This group will receive the routine standard diabetes care.

INTERVENTIONS:
Other: Weight Achievement and Intensive Treatment (Why WAIT) — Weight Achievement and Intensive Treatment (Why WAIT) is a 12 -week multidisciplinary program for weight control and intensive diabetes management designed by the Joslin Diabetes Center for application in a multidisciplinary diabetes practice environment. Participants will be enrolled in a 12-week multidisciplinary intensive weight management including diet, exercise, behavioral and educational support. Participants will be enrolled in cohorts of 10-15 participants to encourage group interaction and support. Subjects will choose to come to the Joslin clinic every Tuesday or Wednesday evening for 2 hours. Participants will exercise for an hour and will attend a didactic session in the areas of nutrition, exercise and behavioral modifications.
  Arms: Intensive Treatment (Why WAIT)

SUMMARY:
The purpose of this study is to find out the impact of improving diabetes control through weight reduction and lifestyle changes on a common diabetes complication called peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion of Intervention group:

1. Men and Women with established Diabetes.
2. BMI between 30-45 Kg/m2
3. Age: 18-75 years old.
4. Enrolled in the Why WAIT program
5. Diabetes duration of at least 5 years
6. Hb A1C of 6.5% or higher

Inclusion of controls:

1. Men and Women with established Diabetes.
2. BMI between 30-45 Kg/m2
3. Age: 18-75 years old.
4. Diabetes duration of at least 5 years
5. Hb A1C of 6.5% or higher

Exclusion Criteria:

1. Anatomic changes that preclude the measurement of the nerve conduction: foot deformities, open skin injuries/ulcers, amputations and placement of surgical plates and screws in the ankle and lower leg (tibial) area.
2. Severe diabetic peripheral neuropathy as defined clinically.
3. Severe peripheral vascular disease e.g absent dorsalis pedis pulsation.
4. Recent weight loss/gain (10 pounds) during the past six months.
5. Neuropathy due to other causes other than diabetes: Alcohol abuse, Liver/Renal disease, Toxic exposure, Inflammatory Disease, Nutritional and Vitamin deficiencies.
6. Individuals with cardiac pacemakers.
7. Women who are Pregnant or who think they might be pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Sural nerve conduction velocity | Baseline, at 3 months, at 6 months, at 12 months
  The NCstat DPNCheck device(an FDA approved device) measures the sural nerve conduction velocity. The sural nerve conduction velocity is the gold standard in assessing diabetic peripheral neuropathy.

SECONDARY OUTCOMES:
Change in Sural Nerve Amplitude potential | Baseline, at 3 months, at 6 months, at 12 months
  The NCstat DPNCheck device(an FDA approved device) measures the sural nerve Amplitude potential. The sural nerve is the gold standard in assessing diabetic peripheral neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Hamdy, MD., PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States